CLINICAL TRIAL: NCT03592121
Title: Study to Investigate the Effect of AB-101 in Breast Cancer Survivors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJ-101-RCT-001
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Sexual Dysfunction; Sexual Arousal Disorder; Sexual Dysfunction, Physiological; Breast Cancer; Nipple Disorder; Neuropathy; Cancer of Breast
Keywords: Nipple Neuropathy, Cancer Survivor
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Breast Neoplasms | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB-101 (Experimental): Apply to both nipple/areola regions approximately 1 hour prior to sexual activity
  Interventions: Drug: AB-101
- Placebo (Placebo Comparator): Apply to both nipple/areola regions approximately 1 hour prior to sexual activity
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AB-101 — Apply approximately 1 hour prior to sexual activity
  Other Names: Phenylephrine
  Arms: AB-101
Drug: Placebo — Apply approximately 1 hour prior to sexual activity
  Other Names: Vehicle Solution
  Arms: Placebo

SUMMARY:
The purpose of this research study is to investigate the possibility that a topical drug could restore nipple sensitivity and improve sexual quality of life in breast cancer survivors.

DETAILED DESCRIPTION:
Approximately, 80% of breast cancer survivors undergoing will suffer from a permanent reduced reduction in nipple sensitivity and associated lowerdecrease in sexual quality of life. Currently, there are no treatments for restoring nipple sensitivity and the associatedto improve lower sexual quality of life this condition. It would thus be of great clinical benefit to post breast surgery patients if a provide a new safe and , effective , topical , on-demand, treatment for this condition can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivor
* Age: 18 to 70
* First diagnosed with Stage I or II breast cancer
* Have had breast surgery: nipple sparring mastectomy or lumpectomy
* At least 3 years post surgery
* Nipple neuropathy post breast surgery (change in Llikeart scale >= 3 between pre and post surgery)
* Baseline nipple sensitivity <=5 (likeartLikert scale)
* QoL-BC (>=7)
* Delayed orgasm (CTCAE v4.0) Grade 2
* One of the following: Delayed orgasm (CTCAE v4.0) Grade 2 and/or Vaginal dryness (CTCAE v4.0) Grade 2 or 3
* Able to give informed consent
* Currently in a monogamous heterosexual relationship for at least 12 months
* Sexually active within the last 30 days
* Willing to engage in sexual activity at least once a month during the duration of the study
* Willing to use on a regular basis a web based form system to record sexual events i.e., have access to the Internet
* Willing to use an adequate method of birth control
* Able to comply with the study requirements for 8 consecutive weeks
* Able to give informed consent

Exclusion Criteria:

* Previous adverse event to alpha 1 agonists (oral, nasal, topical, or ocular) or drugs in this class
* Currently pregnant
* Nursing within the last 6 months prior to beginning the study
* History of cardiovascular or cerebrovascular disease, e.g., heart attack, disease of the arteries of the heart, partial heart block, rapid ventricular heartbeat, slow heartbeat, chronic heart failure, severe hardening of the arteries, blood clot in an artery
* Actively being treated for breast cancer
* Changes in chronic medication for oncology, cardiology, or endocrinology in past 12 months
* Uncontrolled or severe hypertension
* Decreased oxygen in the tissues or blood
* Active inflammation of the liver
* Acute inflammation of the pancreas
* Overactive thyroid gland
* Acidosis
* Diabetes
* Spinal cord injury
* Nipple dermatitis
* Regional complex pain syndrome
* Use of any hypertensive drugs
* Use of MAO inhibitors
* Subjects assigned to interventional drug arm and failed to report an increase >=2 from baseline in nipple sensitivity (likert scale) during phase I
* In partners: sexual dysfunction or erectile dysfunction
* Currently enrolled in any other medical study or has been enrolled in any medical study in the past 30 days
* Nipple dermatitis
* Regional complex pain syndrome
* Unable to provide consent or make allotted clinical visits

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Breast Cancer Survivors
Enrollment: 3 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krychman, MD, Principal Investigator — Southern CA Center for Sexual Health and Survivorship Medicine
Locations (1):
- Southern CA Center for Sexual Health and Survivorship Medicine, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AB-101 | Placebo
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We were unable to recruit a sufficient number of subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | AB-101 | Placebo | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3
Delayed Orgasm Grade (CTCAE v4.0) [Mean (Standard Deviation); unit: Grade] — CTCAE v4.0 is the NIH Common Terminology of Adverse Events v4.0
  Delayed Orgasm is defined as: A disorder characterized by sexual dysfunction characterized by a delay in climax.
  This is a binary grading system:
  Grade 0:Delay in achieving orgasm not adversely affecting relationship Grade 1:Delay in achieving orgasm adversely affecting relationship
  Grade | 0.67 (0.58) |  | 0.67 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change in Delayed Orgasm Grade
Description: Change in Delayed Orgasm Grade (CTCAE v4.0 - Common Terminology of Adverse Events) CTCAE v4.0 is the NIH Common Terminology of Adverse Events v4.0
  Delayed Orgasm is defined as: A disorder characterized by sexual dysfunction characterized by a delay in climax.
  This is a binary grading system:
  Grade 0:Delay in achieving orgasm not adversely affecting relationship Grade 1:Delay in achieving orgasm adversely affecting relationship
Time Frame: [baseline, week 8]
Population: We were unable to recruit a sufficient number of subjects.
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | AB-101 | Placebo
Number analyzed (Participants) | 3 | 0
Grade | -0.33 (0.58) |

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The topical product is used in OTC medications.
Arm/Group | AB-101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03592121/Prot_SAP_000.pdf